CLINICAL TRIAL: NCT07330219
Title: The Effect of Fully Immersive Virtual Reality Technology Combined With Psychological and Behavioral Intervention on Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongren Hongxin Kangxin Traditional Chinese Medicine Hospital, Guizhou Province (Other)
Responsible Party: Principal Investigator, lining, Principal Investigator, Tongren Hongxin Kangxin Traditional Chinese Medicine Hospital, Guizhou Province
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1-1
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fully Immersive Virtual Reality Combined With Psychological and Behavioral Intervention (Experimental): Participants receive fully immersive virtual reality (FIVR) training combined with standard psychological and behavioral intervention (PBI). The intervention lasts for 12 weeks. FIVR is delivered 3-5 times per week in addition to routine PBI.
  Interventions: Behavioral: Fully Immersive Virtual Reality Training; Behavioral: Psychological and Behavioral Intervention
- Psychological and Behavioral Intervention Only (Active Comparator): Participants receive standard psychological and behavioral intervention (PBI) alone for 12 weeks, including language training, sensory integration training, group activities, individualized training, family-based training, and psychological support.
  Interventions: Behavioral: Psychological and Behavioral Intervention

INTERVENTIONS:
Behavioral: Fully Immersive Virtual Reality Training — Fully immersive virtual reality (FIVR) training is delivered using head-mounted display devices. The training includes structured virtual scenarios targeting social interaction, communication skills, and sensory regulation. Each session lasts 20-60 minutes, delivered 3-5 times per week for 12 weeks, with individualized adjustment based on participant tolerance and performance.
  Arms: Fully Immersive Virtual Reality Combined With Psychological and Behavioral Intervention
Behavioral: Psychological and Behavioral Intervention — Psychological and behavioral intervention (PBI) includes language training, sensory integration training, group-based activities, individualized behavioral training, family-based training, and psychological support. Sessions are conducted multiple times per week over a 12-week period according to a standardized rehabilitation protocol.

SUMMARY:
To explore the effects of immersive virtual reality technology combined with psychological and behavioral intervention on children with autism. Methods: A retrospective study was conducted on the clinical data of 120 children with autism admitted to our hospital from January 2024 to October 2024. 58 children received psychological and behavioral intervention alone (control group), while 62 children received psychological and behavioral intervention combined with immersive virtual reality technology (study group). Disease severity (CARS),

DETAILED DESCRIPTION:
This is a single-center, retrospective interventional study evaluating the effects of fully immersive virtual reality combined with psychological and behavioral intervention in children with autism spectrum disorder. Clinical data were retrospectively collected from February 2024 to October 2024. Outcomes were assessed using standardized behavioral and developmental scales.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism spectrum disorder (ASD) according to DSM-5 criteria;
* Age between 2 and 12 years;
* Complete clinical and assessment data available.

Exclusion Criteria:

* Diagnosis of schizophrenia or other psychotic disorders;
* Severe intellectual disability preventing completion of assessments;
* History of epilepsy or uncontrolled seizure disorders;
* Significant visual or auditory impairment;
* History of intracranial surgery or implantation of metallic foreign bodies.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Childhood Autism Rating Scale (CARS) Total Score | Baseline and 12 weeks after initiation of intervention
  The Childhood Autism Rating Scale (CARS) is a clinician-rated assessment consisting of 15 items, each scored from 1 to 4, with a total score range from 15 to 60.
  Higher scores indicate more severe autism-related symptoms (worse outcome). The outcome is defined as the change in total CARS score from baseline to the end of the 12-week intervention period.

SECONDARY OUTCOMES:
Change in Aberrant Behavior Checklist (ABC) Total Score | Baseline and 12 weeks
  The Aberrant Behavior Checklist (ABC) is a standardized caregiver-rated scale assessing problem behaviors in children with autism spectrum disorder across five domains.
  The total score ranges from 0 to 158, with higher scores indicating more severe behavioral problems (worse outcome).
  The outcome is defined as the change in ABC total score from baseline to 12 weeks.
Change in Psychoeducational Profile-Third Edition (PEP-3) Total Score | Baseline and 12 weeks
  The Psychoeducational Profile-Third Edition (PEP-3) is a standardized developmental assessment evaluating cognitive, language, and adaptive functioning in children with autism spectrum disorder.
  Higher scores indicate better developmental functioning (better outcome). The outcome is defined as the change in PEP-3 total score from baseline to 12 weeks.
Parental Satisfaction With Intervention | 12 weeks
  Parental satisfaction with the intervention is assessed using the Newcastle Satisfaction with Nursing Scales (NSNS).
  The scale measures satisfaction across multiple domains, with higher scores indicating greater satisfaction (better outcome).
  Overall satisfaction is assessed at the end of the 12-week intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Hongxinkang New Traditional Chinese Medicine Hospital, Tongren, Tongren, Guizhou, China

REFERENCES:
- [Result] Li N, Tian M, Yang Y, Liu Z, Sun L, Li B. The effect of fully immersive virtual reality technology combined with psychological and behavioral intervention on autism spectrum disorder. BMC Psychol. 2025 Oct 9;13(1):1120. doi: 10.1186/s40359-025-03460-y. PMID 41068944